CLINICAL TRIAL: NCT01929967
Title: Defining Immunodeficiency in Heterotaxy Syndrome: Pilot Study Data
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Litron Laboratories (Industry)
Responsible Party: Principal Investigator, Terence Prendiville, Pediatric Cardiology Fellow, Boston Children's Hospital
Other Study IDs: IRB-P00007001
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Heterotaxy Syndrome
Keywords: Heterotaxy syndrome; Asplenia; Polysplenia
MeSH Terms: conditions — Heterotaxy Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heterotaxy syndrome: Patients with a diagnosis of heterotaxy syndrome, as objectively defined by visceral heterotaxy (malrotation, interrupted inferior vena cava) with either documented polysplenia or asplenia by radiological imaging

SUMMARY:
The investigators aim with this study is to investigate the mechanisms of immune deficiency in patients with heterotaxy syndrome through the use of novel biomarkers and a prospective questionnaire survey documenting the burden of infectious sequelae following enrollment. It is known that patients with under-active spleens (functional asplenia or hyposplenia) secondary to other (non-cardiac) conditions such as Sickle Cell Disease or Inflammatory Bowel Disease have a characteristic paucity of a B cell sub-class known as IgM memory B cell. This specific sub-class of B cell normally matures in the spleen and in those with an improperly functioning spleen a significant deficiency of this B cell class is seen on flow cytometry.

Similarly, these same patients are noted to have increased amounts of 'junk' DNA / nuclear remnant in their red cells. This is seen on microscopy as a dark particle inside the red cell and is termed a Howell Jolly Body (normally less than 2% of red cells have these dark particles present). Part of a functioning spleen's normal task is to rid the blood of red cells that contain nuclear remnants and an under-active spleen gets behind on this task with a build-up of Howell Jolly Bodies in red cells present in the bloodstream. Flow cytometry can very quickly and accurately quantify Howell Jolly Bodies as well as IgM memory B cells from a small (~1.5cc) sample of blood. Normal IgM memory B cell ranges are known for healthy children from infancy onwards allowing interpretation of results against normative data ranges.

The investigators aim to enroll 10 patients in this pilot study who have a diagnosis of heterotaxy syndrome (both asplenia and polysplenia) and to prospectively follow them after obtaining the initial biomarker sample. The family will be contacted once every two weeks for a period of 12 weeks and asked a series of simple questions taking approximately 5 minutes on any recent infectious sequelae or symptoms. The questions will elucidate history of minor illness such as low-grade fever or cough to more significant events such as admission for in-patient antibiotic therapy of bacterial sepsis. Ultimately, with this pilot study, the investigators hope to obtain sufficient data to support funding applications for a larger, multi-center trial that will allow us to develop biomarker thresholds for future risk of sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heterotaxy syndrome, as objectively defined by visceral heterotaxy (malrotation, interrupted inferior vena cava) with either documented polysplenia or asplenia by radiological imaging.
* 0-12 years old.

Exclusion Criteria:

* Other known immunodeficiency or hyposplenic states (22q11, hypogammaglobulinemia, sickle hemoglobinopathy, liver cirrhosis or portal hypertension, organ transplantation, Fanconi syndrome, HIV or AIDS, chronic corticosteroid use, cancer, chemotherapy or other immunomodulating drug exposure, Addison's disease or pan-hypopituitarism, surgical splenectomy).
* Red blood cell transfusion within the last 90 days as the donated red blood cells may interfere with calculation of the subject's Howell Jolly Body count. Patient enrollment will be deferred until 90 days has elapsed, assuming other eligibility requirements are met.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with a diagnosis of heterotaxy syndrome from inpatient and outpatient Cardiology settings at Boston Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Howell Jolly Body quantification | At time of recruitment
IgM Memory B Cell quantification | At time of recruitment

SECONDARY OUTCOMES:
Results of phone questionnaire of parents documenting infectious symptoms and sequelae | Once every 2 weeks for 12 weeks following enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Terence Prendiville, MB BCh BAO, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States